CLINICAL TRIAL: NCT07039110
Title: The Real-World Impact of Risankizumab on the Quality of Life and Cumulative Life Course Impairment (CLCI) in Patients With Moderate-to-Severe Plaque Psoriasis (DREAM)
Brief Title: Study to Assess Change in Quality of Life of Risankizumab Treatment in Adult Participants With Moderate-to-Severe Plaque Psoriasis
Acronym: DREAM
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-187
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Moderate to Severe Plaque Psoriasis; Risankizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Risankizumab: Participants will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
Psoriasis is a chronic, systemic, inflammatory disease in which skin cells build up and develop thick, red and white scaly patches on the skin. This study will assess the change in quality of life of risankizumab treatment in adult participants with moderate to severe plaque psoriasis real-world clinical practice.

Risankizumab is an approved drug for treating participants with Psoriasis. Approximately 700 participants who are prescribed risankizumab by their physician in accordance with local label will be enrolled in approximately 70 sites worldwide.

Participants will receive risankizumab as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 2.5 years.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a Confirmed diagnosis of moderate-to-severe plaque psoriasis with or without joint involvement according to the treating physician's clinical judgment, prior to time of enrollment.
* Treatment with risankizumab is indicated per summary of product characteristics (SmPC) or local label and local prescribing/treatment guidelines.
* Decision to treat with risankizumab is made prior to and independently of study participation.

Exclusion Criteria:

* History of a sleep disorder diagnosis which the patient is currently being treated for.
* Current or recent (within the last 30 days) participation in an interventional clinical trial or an observational study.
* Currently receiving other biologic treatments and/or small molecules including Janus kinase (JAK) inhibitors, tyrosine kinase 2 (TYK2) inhibitors, and phosphodiesterase 4 (PDE4) inhibitors for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate to severe plaque psoriasis who are prescribed risankizumab by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving a Dermatology Life Quality Index (DLQI) score of 0 or 1 | At 12 months
  DLQI (Dermatology Life Quality Index) assesses symptoms and impacts of dermatologic diseases on quality of life. DLQI scores range from 0 (no at all) to 1 (a little).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (50):
- Canada (17):
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 276688, Edmonton, Alberta
  - Winnipeg Clinic /ID# 276751, Winnipeg, Manitoba
  - Wiseman Dermatology Research /ID# 276847, Winnipeg, Manitoba
  - Cca Medical Research /ID# 276944, Ajax, Ontario
  - Quinte dermatology /ID# 277497, Belleville, Ontario
  - Dermatrials Research /ID# 276714, Hamilton, Ontario
  - Lovegrove Dermatology /ID# 276797, London, Ontario
  - Lynderm Research Inc /ID# 276755, Markham, Ontario
  - Rejuvenation Dermatology Clinic Oakville /ID# 277492, Oakville, Ontario
  - JRB Research inc. /ID# 277730, Ottawa, Ontario
  - Factor Dermatology /ID# 278610, Ottawa, Ontario
  - SKiN Centre for Dermatology /ID# 277594, Peterborough, Ontario
  - Eternal Springtime Dermatology /ID# 278598, Thunder Bay, Ontario
  - North York Research Inc /ID# 276835, Toronto, Ontario
  - Toronto Dermatology Centre /ID# 276846, Toronto, Ontario
  - Centre for Medical and Surgical Dermatology /ID# 278775, Whitby, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 276687, Saint-Jérôme, Quebec
- Czechia (4):
  - Nemocnice Na Bulovce /ID# 275540, Prague, Central Bohemia
  - Dermafit Centrum /ID# 275897, Pilsen, Plzeň Region
  - Dermamedest /ID# 275898, Prague, Praha 2
  - Nemocnice Ceske Budejovice /ID# 275541, České Budějovice
- France (3):
  - Centre Hospitalier de Niort Georges Renon /ID# 279604, Niort, Deux-Sevres
  - Dr. Rima Mohty /ID# 279951, Beauvais, Oise
  - Hôpitaux Drôme Nord - Romans /ID# 278109, Romans-sur-Isère
- Germany (6):
  - Dr. med. Moritz Huber und Dr. med. Martin Heister /ID# 277627, Friedrichshafen, Baden-Wurttemberg
  - Dermakulm /Id# 277864, Kulmbach, Bavaria
  - Dermatologie Moelln Praxis Dr. Bodo Segert /ID# 277628, Mölln, Schleswig-Holstein
  - Private Practice - Dr. Mario Pawlak /ID# 277465, Heilbad Heiligenstadt
  - Hautarztpraxis Dr. Med. Ulrike Wiemers / Dr. Med. Franca Wiemers /ID# 277821, Leipzig
  - Hautarztpraxis Schwelm /ID# 277464, Schwelm
- Greece (8):
  - General Hospital Andreas Syggros /ID# 276826, Athens, Attica
  - General Hospital Andreas Syggros /ID# 279246, Athens, Attica
  - Tzaneio Prefecture General Hospital of Piraeus /ID# 276532, Piraeus, Attica
  - Asklipieio General Hospital of Voula /ID# 278235, Voula, Attica
  - The University Hospital of Larissa /ID# 276576, Larissa, Larisa
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 276488, Thessaloniki
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 276489, Thessaloniki
  - Papageorgiou General Hospital /ID# 276487, Thessaloniki
- Italy (2):
  - ASL 1 Abruzzo - Ospedale regionale San Salvatore /ID# 277341, L’Aquila, L Aquila
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 278080, Rome, Roma
- Japan (9):
  - Hokkaido University Hospital /ID# 278260, Sapporo, Hokkaido
  - Hosui General Medical Clinic /ID# 279520, Sapporo, Hokkaido
  - Kagoshima University Hospital /ID# 278514, Kagoshima, Kagoshima-ken
  - Yokohama City University Hospital /ID# 278257, Yokohama, Kanagawa
  - Kawasaki Medical School Hospital /ID# 278259, Kurashiki, Okayama-ken
  - Kindai University Hospital /ID# 278258, Sakai-shi, Osaka
  - Juntendo University Hospital /ID# 278495, Bunkyo-ku, Tokyo
  - Fukuoka University Hospital /ID# 278600, Fukuoka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 278434, Osaka
- Hospital General Universitario Santa María Del Rosell /ID# 277894, Cartagena, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-187